CLINICAL TRIAL: NCT06392321
Title: Dexmedetomidine Versus Fentanyl as an Adjuvant to Single Low Dose Spinal Anesthesia in Controlling Labor Pain: a Randomized Controlled Study
Brief Title: Dexmedetomidine vs Fentanyl in Controlling Labor Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ismail Mohamed Abdelgawad Ahmed, Dr, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: controlling labor pain
Record Dates: First submitted 2024-04-26; First posted 2024-04-30 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Labor Pain
Keywords: Dexmedetomidine; Fentanyl; intrathecal; labor pain
MeSH Terms: conditions — Labor Pain | interventions — Fentanyl; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fentanyl (Active Comparator): Bupivacaine 3,75 mg + 2.5 ml saline added to fentanyl 20 microgram + 2.3 ml saline
  Interventions: Drug: Fentanyl
- Dexmedetomidine (Active Comparator): Bupivacaine 3,75 mg + 2.5 ml saline added to dexmedetomedine 5 microgram + 2.3 ml saline
  Interventions: Drug: Dexmedetomidine
- control (No Intervention): Bupivacaine 3,75 mg + 2.5 ml saline

INTERVENTIONS:
Drug: Fentanyl — comparison between bupivacaine, bupivacaine and fentanyl.
  Arms: Fentanyl
Drug: Dexmedetomidine — comparison between bupivacaine, bupivacaine and dexmedetomidine..
  Arms: Dexmedetomidine

SUMMARY:
As most woman experience agonizing pain throughout vaginal labor. Adjuvants were added to intrathecal bupivacaine aiming to improve the quality of analgesia. This study aimed to assess the efficacy and outcome of intrathecal dexmedetomidine and fentanyl in controlling pain during delivery.

DETAILED DESCRIPTION:
Throughout vaginal deliveries, many women suffered from pain. providing suitable analgesia is crucial (Lupu et al., 2023). Spinal anesthesia can provide pain management (Parikh et al., 2018).

Various types of analgesics can be combined to get the needed duration of perioperative analgesia. Dexmedetomidine has been used with effective pain management outcomes (Shrestha et al., 2023). Fentanyl can help pain relief in short duration procedures (Show et al., 2022).

ELIGIBILITY:
Inclusion Criteria:

* women planned for spontaneous vaginal delivery.

Exclusion Criteria:

* cardiac, liver or kidney disease, allergy to local anesthetics or the studied drugs, any contraindication of regional anesthesia and intrauterine growth retardation or fetal compromise.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
efficacy of intrathecal dexmedetomidine | 120 minutes
  VAS

SECONDARY OUTCOMES:
patient satisfaction | 2 hours
  satisfaction score
mother's outocme | 1 and 5 minutes
  APGAR

CONTACTS AND LOCATIONS:
Locations (1):
- Al Azhar University, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: No
IPD are planned to be coded for privacy protection.

REFERENCES:
- [Background] Lupu VV, Miron IC, Raileanu AA, Starcea IM, Lupu A, Tarca E, Mocanu A, Buga AML, Lupu V, Fotea S. Difficulties in Adaptation of the Mother and Newborn via Cesarean Section versus Natural Birth-A Narrative Review. Life (Basel). 2023 Jan 21;13(2):300. doi: 10.3390/life13020300. PMID 36836657
- [Background] Parikh KS, Seetharamaiah S. Approach to failed spinal anaesthesia for caesarean section. Indian J Anaesth. 2018 Sep;62(9):691-697. doi: 10.4103/ija.IJA_457_18. PMID 30237594
- [Background] Shrestha IK, Chalise R, Poudel S, Regmi A, Ghimire A, Khadka B, Khanal K. Neostigmine and atropine as a treatment for postdural puncture headache after spinal anesthesia in cesarean section: A case report. Clin Case Rep. 2023 Nov 2;11(11):e8132. doi: 10.1002/ccr3.8132. eCollection 2023 Nov. PMID 37927977
- [Background] Show KL, Ngamjarus C, Kongwattanakul K, Rattanakanokchai S, Duangkum C, Bohren MA, Betran AP, Somjit M, Win WYH, Lumbiganon P. Fentanyl for labour pain management: a scoping review. BMC Pregnancy Childbirth. 2022 Nov 17;22(1):846. doi: 10.1186/s12884-022-05169-x. PMID 36397024